CLINICAL TRIAL: NCT02848560
Title: Validation of MRI as a Sensitive Tool to Longitudinally Monitor CF Lung Disease Progression and Response to CFTR Modulator Therapy in Young Children With CF
Brief Title: Monitoring Response to Orkambi in Cystic Fibrosis Lung Disease by Inhaled Xenon MRI
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jason Woods, PhD, Children's Hospital Medical Center, Cincinnati
Other Study IDs: CINOO1-CF Orkambi and Xe MRI; 1R01HL131012-01A1 (NIH)
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; orkambi; 129Xe MRI; hyperpolarized xenon; LCI; CFTR modulator therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment: Observation of lung changes over time by hyperpolarized xenon MRI on CF patients homozygous for F508del CFTR mutation as they age into the FDA approved treatment window for the CFTR modulator orkambi. Subjects will be observed at 2 time points before starting clinically prescribed treatment (orkambi) and 2 time points while on orkambi.
  Interventions: Drug: Hyperpolarized Xenon
- Control: Observation of lung changes over time by hyperpolarized xenon MRI on CF patients heterozygous for F508del CFTR mutation at similar timepoints to treatment group. Control subjects are not be eligible to be clinically prescribed orkambi based on FDA approval.
  Interventions: Drug: Hyperpolarized Xenon

INTERVENTIONS:
Drug: Hyperpolarized Xenon — Inhaled contrast for MRI occurring at each of 4 visits.
  Other Names: 129Xe

SUMMARY:
This is an observational study for children with Cystic Fibrosis (CF) who are eligible based on their CF gene type. One group will be called the treatment group because they have the gene type (homozygous F508del) that makes them clinically eligible through their CF care provider to begin treatment with the new FDA approved CF drug called orkambi. For the control group, children will be enrolled who have a similar CF gene type (heterozygous F508del) but are not eligible to be prescribed orkambi.

The two groups will be followed for four visits over about 3 to 4 years to observe changes in the lungs. Methods to measure the changes in lung disease will include:

MRI with non-FDA approved inhaled xenon gas to take detailed images of the lungs, Pulmonary Function Tests (PFT), Lung Clearance Index (LCI), Baseline CT image of the lungs if not ordered as part of usual clinical care.

The first two visits will be done before starting clinical treatment with orkambi and will be a minimum of 28 days apart and up to 18 months. The third visit will be scheduled about 3 months after starting orkambi and the fourth visit about 18 months later. For the control group, the timing of visits will be similar to treatment group and visits may be scheduled around annual CF care visits.

DETAILED DESCRIPTION:
This is a controlled observational longitudinal study designed to capture Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) modulator therapy naive Cystic Fibrosis (CF) subjects with F508del(+/+) mutations before they age into the FDA approved treatment window for the CFTR modulator orkambi (ivacaftor/lumacaftor). These subjects will be compared to disease controls. The treatment group will be observed twice (at least 28 days apart and up to 18 months) before clinically starting orkambi and observed twice (at about 3 months and about 18 months) after clinically starting orkambi .

This study takes advantage of the timely development of Ultrashort Echo Time Magnetic Resonance Imaging (UTE MRI), Hyperpolarized Xenon (129Xe) MRI, Lung Clearance Index (LCI), and the approval of F508del CFTR-directed CF therapy in children. The proposal will:

i) validate the emerging biomarker (UTE MRI) within CF children independent of genotype, ii) define the trajectory of UTE MRI and forced expiratory volume in 1 second (FEV1) changes before and after initiating orkambi therapy compared with age-matched CF controls, and iii) determine the relationships between regional structural abnormalities (UTE MRI) and regional (129Xe MRI) and global (LCI) functional measures of ventilation. Results will establish MRI as a sensitive lung imaging tool that is translatable to all CF centers and can be applied throughout the lifespan of CF patients.

CF patients with one or two copies of the F508del CFTR mutation who are 6-12 years old will undergo UTE MRI soon after a clinical computerized tomography (CT) scan, with disease quantification using an established scoring system for both modalities. Quantitative imaging data and LCI will be compared with spirometry (gold standard for CF lung disease) and clinical predictors of disease progression.

The F508del(+/+) patient cohort will differ genotypically from the control cohort (F508del[+/-]). All patients in the F508del(+/-) cohort will be pancreatic insufficient and also have a nonfunctional second allele (Class I or II mutation, not candidates for modulator therapy). These two cohorts are phenotypically indistinguishable without modulator treatment, and therefore the untreated cohort will serve as an ideal age and time-matched control group for the F508del(+/+) subjects who clinically initiate orkambi.

Disease trajectories in the two groups, as quantified by changes in pulmonary UTE MRI, will be compared with FEV1. MRI analysis will include quantitative and reader-based "Brody" scoring for the whole lung, lung lobes, and for subcategories of the Brody scoring system (in particular bronchiectasis, bronchial wall thickening, and mucus plugging).

The longitudinal study will capture both cohorts at their scheduled annual CF visits when possible over about 4 years with modifications to the timeline for the treatment group based on when they are clinically scheduled to begin orkambi treatment.

As FDA approved indications for orkambi change, subjects in the F508del(+/+) cohort will become candidates for modulators prior to their 12th birthday. The FDA is currently reviewing for approval in Fall 2016 to lower the prescribing age to 6 years and the investigators will be enrolling to meet the changes at that time.

ELIGIBILITY:
Inclusion Criteria:

Treatment group:

* male or female between the ages of 6 through 12 years at enrollment
* two copies of the F508del CFTR mutation
* anticipated to be a candidate for treatment with orkambi

Control group:

* male or female between the ages of 6 through 12 years at enrollment
* two non-functional CFTR mutations with one of them being F508del CFTR mutation
* not eligible for CFTR modulation therapy

Exclusion Criteria:

* FEV1 percent predicted of <60%
* standard MRI exclusions (metal implants, claustrophobia)
* pregnancy

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cystic Fibrosis patients naïve to orkambi and with either homozygous F508del CFTR mutation or heterozygous F508del CFTR mutation and pancreatic insufficient.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Hyperpolarized 129Xe MRI Image Analysis | Visit 4 (year 3)
  Lung defect calculations (total and lobar defect percentages) will be performed by evaluating the percentage of voxels with signals below a threshold value of 60% of the total lung mean signal.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Woods, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
MRI results will be shared with treating CF physicians to support clinical decisions.